CLINICAL TRIAL: NCT01526668
Title: A Randomized Study Comparing Four Different Postoperative Follow-up Strategies for Improved Postoperative Recovery After Benign Hysterectomy
Brief Title: Follow-up Strategies for Improved Postoperative Recovery After Benign Hysterectomy
Acronym: POSTHYSTREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Preben Kjolhede, MD, professor, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POSTHYSTREC
Record Dates: First submitted 2012-01-27; First posted 2012-02-06 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Hysterectomy; Genital Diseases, Female; Pain
Keywords: Benign gynecological disease; Surgery; Postoperative follow-up strategy; Pain threshold; Chronic pelvic pain; [E04.950.300.399]; [C13.351.500]; [F02.463.593.710.560]; [N02.421.585.722.700]; Postoperative Care
MeSH Terms: conditions — Genital Diseases, Female; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No contact after discharge (Active Comparator): In Arm A: The patient do not have planned contacts with the study nurse or doctor after discharge. All patients are seen by the study nurse six weeks postoperatively.
  Interventions: Behavioral: No contact after discharge
- Single telephone contact (Active Comparator): In Arm B: The patient has one planned telephone contact with the study nurse the day after discharge. All patients are seen by the study nurse six weeks postoperatively.
  Interventions: Behavioral: Follow-up strategy
- Telephone contacts regularly (Active Comparator): In Arm C: The patient has planned telephone contacts with the study nurse the day after discharge and then once weekly until the six weeks follow-up visit postoperatively.
  Interventions: Behavioral: Follow-up strategy
- Telephone contact using CBT-inspired strategy (Active Comparator): In Arm C: The patient has planned telephone contacts with the study nurse the day after discharge and then once weekly until the six weeks follow-up visit postoperatively. At these telephone contacts the study nurse uses a cognitive behavior therapy (CBT)-inspired strategy in counselling and support.
  Interventions: Behavioral: Follow-up strategy

INTERVENTIONS:
Behavioral: Follow-up strategy — Comparison of different follow-up strategies
  Arms: Single telephone contact; Telephone contact using CBT-inspired strategy; Telephone contacts regularly
Behavioral: No contact after discharge
  Arms: No contact after discharge

SUMMARY:
The purpose of the study is to investigate the effect of four different follow-up strategies on postoperative recovery following vaginal or abdominal hysterectomy for benign conditions. Furthermore the investigators aim to examine associations between preoperative thresholds for pain (thermal and pressure) and postoperative pain and development of chronic pelvic pain after benign hysterectomy.

DETAILED DESCRIPTION:
Contact sponsor if detailed information is requested.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 60 years of age.
* Women who are scheduled for vaginal or abdominal total or subtotal hysterectomy for benign gynecological diseases (including cervical dysplasia).
* Women who understand and speak Swedish fluently.
* Women who gives signed informed consent to participate in the study.
* Women who have access to a telephone and/or internet.

Exclusion Criteria:

* Women where the hysterectomy is carried out in association with surgery for genital prolapse
* Women with genital malignancies (does not include cervical dysplasia).
* Women where the operation is planned or expected to comprise more than the hysterectomy with or without unilateral salpingooophorectomy and appendectomy en passant.
* Women with previous bilateral salpingooophorectomy.
* Women who are physically disabled to a degree so that mobilization postoperatively cannot be expected as for a normal individual.
* Women who are mentally disabled to a degree so she cannot complete the forms in the study or understand the tenor of the participation or it is considered doubtful from an ethical point of view to participate.
* Women with psychiatric disease or is on medication for severe psychiatric disease so that the physician consider participation in the study unsuitable.
* Women with current drug or alcohol abuse.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 525 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Quality of life as measured by the EQ-5D health index | Six weeks
  The Euroqol questionnaire form (EQ-5D) are used for assessing the quality of life. Assessments preoperatively, once daily the first week postoperatively and then once weekly for additional five weeks.
Quality of life as measured by the SF-36 sub scale scores | Six weeks
  The Short-Form 36 (SF-36) are used for assessing the quality of life. Assessments preoperatively, and after six weeks

SECONDARY OUTCOMES:
Postoperative symptoms | Six weeks
  Selfreported symptoms in the Swedish Postoperative Symptom Questionnaire. Assessments preoperatively, once daily the first week postoperatively and then once weekly for additional five weeks.
Consumption of analgesic | Six weeks
  Total amount of opioids and non-opioids from surgery to six weeks postoperatively
Complications related to operation | Six weeks
  From surgery to six weeks postoperatively
Health economy | Up to 1 years
  Direct and indirect costs, quality adjusted life years (QALYs). From surgery to return to work
Development of chronic pelvic pain | One year
  Development of chronic pelvic pain one year postoperatively among women with no pelvic pain preoperatively
Duration of sick-leave | Up to one year
  Time from day of surgery to return to work at same level as preoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kjolhede, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, 58185 Linkoping, Sweden; Ninnie Borendal Wodlin, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, S-58185 Linkoping, Sweden; Lena Nilsson, MD, PhD, Study Chair — Department of Anesthesiology, University Hospital, S-58185 Linkoping, Sweden; Gunilla Sydsjo, PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, S-58185 Linkoping, Sweden; Gulnara Kassymova, MD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, S-58185 Linkoping, Sweden; Peter Lukas, MD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, S-58185 Linkoping, Sweden; Björn Gerdle, MD, PhD, Study Chair — Pain and Rehabilitation Center, University Hospital, 581 85 Linkoping, Sweden
Locations (5):
- Sweden (5):
  - Department of Obstetrics and Gynecology, Höglandshospital, Eksjö, Jonkopings Län
  - Department of Obstetrics and Gynecology, Ryhov Central Hospital, Jönköping, Jonkopings Län
  - Department of Obstetrics and Gynecology, Värnamo, Jonkopings Län
  - Department of Obstetrics and Gynecology, University Hospital, Linköping, Östergötland County
  - Department of Obstetrics and Gynecology, Vrinnevi Hospital, Norrköping, Östergötland County

REFERENCES:
- [Derived] Kassymova G, Davidson T, Sydsjo G, Wodlin NB, Nilsson L, Kjolhede P. Cost analysis of nurse-lead telephone follow-ups after benign hysterectomy: a randomized, single-blinded, four-arm, controlled multicenter trial. Arch Gynecol Obstet. 2025 Aug;312(2):515-523. doi: 10.1007/s00404-025-08035-1. Epub 2025 May 2. PMID 40314809
- [Derived] Lukas P, Nilsson L, Wodlin NB, Arendt-Nielsen L, Kjolhede P. Changes in spatial bodily pain distribution one year after benign hysterectomy with emphasis on prevalence and risk factors for de novo and persistent pelvic pain- a prospective longitudinal multicenter study. BMC Womens Health. 2024 Dec 20;24(1):644. doi: 10.1186/s12905-024-03474-5. PMID 39707275
- [Derived] Kassymova G, Sydsjo G, Borendal Wodlin N, Nilsson L, Kjolhede P. The Impact of Symptoms of Depression, Anxiety, and Low Stress-Coping Capacity on the Effects of Telephone Follow-Up on Recovery Measures After Hysterectomy. Womens Health Rep (New Rochelle). 2024 Mar 27;5(1):304-318. doi: 10.1089/whr.2023.0045. eCollection 2024. PMID 38558946
- [Derived] Kassymova G, Sydsjo G, Wodlin NB, Nilsson L, Kjolhede P. Effect of nurse-led telephone follow-up on postoperative symptoms and analgesics consumption after benign hysterectomy: a randomized, single-blinded, four-arm, controlled multicenter trial. Arch Gynecol Obstet. 2023 Feb;307(2):459-471. doi: 10.1007/s00404-022-06722-x. Epub 2022 Sep 2. PMID 36050542
- [Derived] Kassymova G, Sydsjo G, Borendal Wodlin N, Nilsson L, Kjolhede P. The Effect of Follow-Up Contact on Recovery After Benign Hysterectomy: A Randomized, Single-Blinded, Four-Arm, Controlled Multicenter Trial. J Womens Health (Larchmt). 2021 Jun;30(6):872-881. doi: 10.1089/jwh.2020.8752. Epub 2020 Nov 24. PMID 33232628